CLINICAL TRIAL: NCT01583959
Title: Randomized Trial of 10 mg Versus 30 mg Per Week of Folic Acid in Combination With Methotrexate in Rheumatoid Arthritis
Brief Title: Study of Different Doses of Folic Acid in Combination With Methotrexate in Rheumatoid Arthritis
Acronym: FOLVARI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Varun Dhir, Assistant Professor, Internal Medicine, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-124
Record Dates: First submitted 2012-03-15; First posted 2012-04-24 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; folic acid; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Folic acid 30 mg per week (Active Comparator): Patients will be administered 5 mg folic acid for 6 days a week, no tablet on the day they take methotrexate (5 mg x 6 days = 30 mg per week)
  Interventions: Drug: Folic Acid
- Folic acid 10 mg (Active Comparator): Patients will be given folic acid 5 mg for two days per week and placebo tablets for four days a week, no tablet on the day they take methotrexate (Folic acid 5mg x 2 days = 10mg per week)
  Interventions: Drug: Folic Acid; Drug: Placebo

INTERVENTIONS:
Drug: Folic Acid — Folic acid tablets 5 mg
Drug: Placebo — Matched placebo to folic acid 5 mg tables, to be given for 4 days a week
  Arms: Folic acid 10 mg

SUMMARY:
Introduction: Methotrexate is the sheet anchor for the treatment of rheumatoid arthritis. Folic acid supplementation is usually given at a dose of 5-30 mg per week to ameliorate adverse effects. Patients at our center are usually on the higher dose. However, it is unclear if higher doses are required, recent international recommendations suggest 5-10 mg per week only.

Objectives: To randomize rheumatoid patients being being started on Methotrexate into 2 groups- one on 5mg for 6 days a week (30mg per week) of folic acid and the other 5 mg twice a week (10 mg per week) for 24weeks. To look at difference in

1. Adverse effects due to methotrexate

   a. Minor adverse effects: By symptom chart

   a. Major adverse effects: Cytopenia (predefined) and transaminitis.
2. Disease activity using Disease activity score 28 joints (3 variable) and functional status by health assessment questionnaire
3. RBC folic acid levels Methodology: Randomised controlled trial, double blinded, placebo controlled. Sample size 50 in each group. One group of patients will receive folic acid 5 mg twice a week with placebo for 4 days and the other group will receive folic acid 5 mg 6 days a week for 24 weeks.

Patients will be administered adverse effects proforma, assessed for having cytopenias and transaminitis (pre defined) and disease activity will be calculated at every visit, ie., in the beginning at then at 8,16 and 24 weeks. In addition will look at the functional status and RBC folate levels at 0 and 24 weeks. Statistical analysis using chi-square test for proportions and t test for continuous variables.

DETAILED DESCRIPTION:
THIS TRIAL WILL INCLUDE NEW RHEUMATOID ARTHRITIS PATIENTS These patients will then be randomized into two groups - one which continues to take the same folic acid dose and one which is shifted to folic acid 10 mg per week.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Patients fulfilling the 1987 American College of Rheumatology Rheumatoid arthritis criteria

Exclusion Criteria:

* Hb less than 8 g per dl or TLC less than 3500 or Platelet less than 1 lac or SGOT or SGPT more than 60 U/L
* Serious concomitant medical illnesses such as cancer, liver or renal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Adverse effects | 24 weeks
  i. Minor: Two Symptom charts: Those AEs related temporally to methotrexate and those not temporally related.
  ii. Major: Hemoglobin (Hb), Platelet, Total leucocyte count or white blood count (TLC), Differential leukocyte count (DLC), Serum glutamic oxaloacetate transaminase (SGOT)/ serum glutamic pyruvate transaminase (SGPT) will be done at 3 months. Patients having Hb≤6, TLC ≤ 3500, Platelet ≤99000, SGOT or SGPT ≥80 IU/L
disease activity | 24 weeks
  Using disease activity score 28 joints 3 variables(DAS 28-3v) : uses evaluation of tender joint count (TJC28), Swollen joint count (SJC28) and the erythrocyte sedimentation rate (ESR) using Westergren method.

SECONDARY OUTCOMES:
RBC folic acid: | 24 weeks
  This will be done by chemiluminescence assay, to compare folic acid levels at baseline and at 24 weeks
Function | 24 weeks
  Look at the function by Indian Health assessment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Varun Dhir, MD, DM, Principal Investigator — PGIMER, Chandigarh, India
Locations (1):
- New OPD, #3035, Level 3, Rheumatology Clinic, Tuesday and Friday, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Dhir V, Sandhu A, Kaur J, Pinto B, Kumar P, Kaur P, Gupta N, Sood A, Sharma A, Sharma S. Comparison of two different folic acid doses with methotrexate--a randomized controlled trial (FOLVARI Study). Arthritis Res Ther. 2015 Jun 11;17(1):156. doi: 10.1186/s13075-015-0668-4. PMID 26063325